CLINICAL TRIAL: NCT04550988
Title: Self-conducted Sonographic Monitoring of the Target Joints in Patients With Severe Haemophilia
Brief Title: Sonography and Haemophilia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Principal Investigator, PD Dr. Andreas Strauß, Specialist in orthopedics and trauma surgery, University Hospital, Bonn
Other Study IDs: POD10816
Record Dates: First submitted 2020-08-25; First posted 2020-09-16 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Sonography; Haemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Feasibility Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with severe haemophilia A or B: * Adult patients (≥ 18 years of age) suffering from severe haemophilia A or B
  * No professional medical background
  * Submitted written consent to participate in the study and to use their study related pseudonymised data
  Interventions: Other: feasibility study

INTERVENTIONS:
Other: feasibility study — The aim of this study is to evaluate the possibility of establishing a patient-based ultrasound monitoring of the knee (representing a target joint accessible with any hand) with a handheld device.

SUMMARY:
The aim of this study is to evaluate the possibility of establishing a patient-based ultrasound monitoring of the knee (representing a target joint accessible with any hand) with a handheld device:

The following questions will be answered:

1. What is necessary for the organisational implementation of a patient-based ultrasound monitoring in patients with haemophilia?
2. Is it possible to train patients with haemophilia to perform sonography of their target joints?
3. Does a patient-based ultrasound monitoring with a handheld device work in a home setting?
4. What is the quality of the patient's self-acquired ultrasound images?
5. Will the test persons be able to distinguish normal findings from (any) pathologic findings?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) suffering from severe haemophilia A or B
* No professional medical background
* Submitted written consent to participate in the study and to use their study related pseudonymized data

Exclusion Criteria:

* Patients suffering from other bleeding diseases
* Participants < 18 years of age
* Participants without written consent
* Professional medical background

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) suffering from severe haemophilia A or B. Haemophilia is an X-linked recessive genetic bleeding disease characterised by absence or deficiency of factor VIII in haemophilia A or factor IX in haemophilia B. This can cause spontaneous bleedings, particularly into joints. Joint bleedings initiate an inflammatory process characterised by chronic synovitis that causes degeneration of the affected joints and results in haemophilic arthropathy
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Landmarks of the Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) protocol - Anterior mid-sagittal ultrasound image | 5 min
  The patients will perform an ultrasound of their left and right knee according to the HEAD-US protocol. The following ultrasonic image is needed: Anterior mid-sagittal ultrasound image.
  Patella, distal femur, suprapatellar recess, suprapatellar fat pad and prefemoral fat pad must be visible.
Landmarks of the Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) protocol - Anterolateral transverse ultrasound image | 5 min
  The patients will perform an ultrasound of their left and right knee according to the HEAD-US protocol. The following ultrasonic image is needed: Anterolateral transverse ultrasound image.
  Patellofemoral joint, lateral parapatellar recess, lateral patellar retinaculum and lateral femoral condyle must be visible.
Landmarks of the Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) protocol - Transverse ultrasound image - Transverse ultrasound image | 5min
  The patients will perform an ultrasound of their left and right knee according to the HEAD-US protocol. The following ultrasonic image is needed: Transverse ultrasound image.
  Medial facets of the trochlea, lateral facets of the trochlea and cartilage must be visible.
Landmarks of the Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) protocol - Coronal ultrasound image | 5 min
  The patients will perform an ultrasound of their left and right knee according to the HEAD-US protocol. The following ultrasonic image is needed: Coronal ultrasound image.
  Medial meniscus, boundaries of the femur, boundaries of the tibia must be visible.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Strauß, PD Dr., Principal Investigator — Medicine of the University of Bonn
Locations (1):
- University Hospital of Bonn, Bonn, Northrhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No
The publication of anonymous patient data is not allowed by informed consent.